CLINICAL TRIAL: NCT04570514
Title: Effects and Mechanism of Adipokines Cardiac Protection in Obese Patients With Acute Myocardial Infarction (AMI) Who Have Undergone Percutaneous Coronary Intervention (PCI).
Brief Title: Optimized Cardioprotection Therapy in Obese Subjects With AMI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, sunddong, Cardiology department, Xijing Hospital
Other Study IDs: OB-AMI
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Acute Myocardial Infarction; Myocardial Reperfusion Injury; Obesity; Adiposis; Heart
Keywords: Adiposis; Obesity; Acute Myocardial Infarction; Percutaneous Coronary Intervention; Left Ventricular Function
MeSH Terms: conditions — Myocardial Reperfusion Injury; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obesity: Patients with Obesity. BMI>=25
  Interventions: Procedure: PCI
- Non-Obesity: Patients without Obesity. BMI<25
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — percutaneous coronary intervention (PCI)

SUMMARY:
The purpose of this study is to investigate the efficacy and mechanism of Adipokines Cardiac Protection in Obese Patients With acute myocardial infarction (AMI) Who Have Undergone Percutaneous Coronary Intervention (PCI).

DETAILED DESCRIPTION:
Adipokines (or adipocytokines) can be defined as a group of more than 600 bioactive molecules made from adipose tissue that acts as paracrine and endocrine hormones. Adipokines are involved in maintaining varieties of processes such as, appetite and satiety, energy expenditure activity, endothelial function, blood pressure, hemostasis, adipogenesis, insulin sensitivity, energy metabolism in insulin-sensitive tissues, fat distribution and insulin secretion in pancreatic β-cells. Adipokines may contribute to reduce scar formation and improve cardiac function in acute myocardial infarction (AMI). Reperfusion therapy such as percutaneous coronary intervention (PCI) should be administered to all eligible patients with AMI symptom onset within the prior 12 hours. However, our previous work showed that obese patients may benefit more from PCI. Thus, the aim of the present study was to investigate the efficacy and mechanism of adipokines cardiac protection for obese and non-obese patients with acute myocardial infarction (AMI) who have undergone PCI.

ELIGIBILITY:
Inclusion Criteria:

age between 20 and 70 years old STEMI and NSTMI according to the WHO definition PCI <12 hours from the onset of symptoms

Exclusion Criteria:

previous myocardial infarction (MI) cardiomyopathy atrial fibrillation or flutter previous heart surgery severe valvular heart disease disease of the hematopoietic system NYHA functional class IV heart failure at baseline severe renal, lung and liver disease cancer

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of AMI were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patient death during the follow up period | 1 year

SECONDARY OUTCOMES:
Left ventricular ejection fraction | 1 year
Myocardial perfusion scores as evaluated by Single-photon emission computed tomography (SPECT) | 1 year
Infarct size as evaluated by Single-photon emission computed tomography (SPECT) | 1 year
Number of target vessel revascularization | 1 year
Angina class according to the canadian cardiovascular society (CCS) classification | 1 year
Scores on the Seattle angina questionnaire | 1 year
six-min walk distance (6MWD) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dongdong Sun, M.D.,Ph.D, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China